



THOMAS DRIVE, LIVERPOOL, L14 3PE Telephone 01512281616

| IRAS I | D: 256927 | | | |
|---|---|---|---|---|
| Centr | e Number: | | | |
| Study | Number: | | | |
| Partic | ipant Identification Nu | mber: | | |
| CONS | ENT FORM | | | |
| contro | of Project: A High-pro<br>olled trial<br>of Researcher: Fatima | | and resistance exercise for cardiac rehab | ilitation: a pilot randomised |
| IVAITIC | or nesearcher, ratima | Terez de Heredia | | Please initial box |
| 1. | | ad the opportunity to consid | ated) for the ler the information, ask questions and have | |
| 2. | • | | d that I am free to withdraw at any time re or legal rights being affected. | |
| 3. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by researchers from Liverpool John Moores University, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | |
| 4. | I agree to audio recor | dings being created for the p | ourpose of this study. | |
| 5. | I agree to gift the research team a sample of my blood for the purpose of this study. | | | |
| 6. | <ol> <li>I understand that the information and samples collected from me will be used to support<br/>other research in the future, and may be shared anonymously with other researchers and that a<br/>samples and data will be destroyed after 10 years.</li> </ol> | | | at all |
| 7. | I agree to my General Practitioner being informed of my participation in the study. I agree to my General Practitioner being involved in the study, including any necessary exchange of information about me between my GP and the research team. | | | |
| 8. | I agree to be contacted by the research team approximately 6-months after completion of the s to be asked further questions about my food and exercise habits. | | | e study |
| 9. | I agree to take part in | | | |
| Name | of Participant | Date | Signature | Participant ID |
| | of Person | Date 1 for researcher site file: 1 to b | Signature | |





THOMAS DRIVE, LIVERPOOL, L14 3PE Telephone 01512281616

taking consent